CLINICAL TRIAL: NCT06589466
Title: Retrospective Review of Preoperative Optimization of Diabetic Patients
Brief Title: Preoperative Optimization of Diabetic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00139994
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Surgery Related Complications Rate
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with diabetes having surgery in Alberta since November 2019: Adults with diabetes having surgery in Alberta since November 2019
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — this study in observational study, no intervention.

SUMMARY:
Diabetic patients, as part of preoperative evaluation, should have glycated hemoglobin (HbA1C) measured. HbA1C provides information on longterm glucose control. There is a suggestion in the literature that elevated A1C levels predict a higher rate of postoperative adverse events, including infections, myocardial infarction, and mortality. It is unclear whether chronic glycemia, as reflected in raised HbA1C level, is the risk factor for adverse perioperative events or whether it is a surrogate measure for poor perioperative glucose management. Conversely, in a retrospective analysis of 431,480 surgeries perioperative glucose was predictive of increased 30-day mortality, but that HbA1C was a less useful predictor of this measure. In our experience of at the University of Alberta Preadmission Clinic there is significant variability with respect to whether diabetic patients have a valid HbA1C measurement i.e. within 3 months of surgery. If a valid measurement is present, there is also considerable variability with respect to diabetes control.

DETAILED DESCRIPTION:
Purpose: The purpose of this study to retrospectively determine the incidence of diabetes in the surgical population and what proportion of diabetic patients have a valid HbA1C. Hypothesis: A valid (measured within 3 months of surgery) HbA1C measurement is frequently missing prior to surgery and when present has a high chance of being higher than normal.

Objectives:

Perform a retrospective analysis of all surgeries in Alberta from November 2019 to the present time looking for the following:

Primary outcomes:

1. Determine the incidence of diabetes in the surgical population and describe the demographics and clinical charcteristics of patients
2. Determine the incidence of valid HbA1C in diabetic patients presenting for surgery
3. Determine long-term diabetes control through assessment of HbA1C values in diabetic patients presenting for surgery

Secondary outcomes:

1. Determine association between HbA1C and post-operative length of stay
2. Determine association between HbA1C and in hospital mortality Design: This study will be a population-based, retrospective observational cohort study. Setting: Alberta Hospitals Participants: Adults with diabetes having surgery in Alberta since November 2019 Descriptive statistics will be tabulated according to HbA1C status and Univariate comparisons of means, medians and proportions will be performed to evaluate the association of independent variables with primary and secondary outcomes. Normally distributed continuous data will be reported as means with standard deviations (SD). Non-normally distributed continuous data will be reported as medians with interquartile ranges (IQR). Categorical variables will be compared using Chi-square test for independence

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Having any surgical procedure at any hospital in Alberta

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Adults having any surgical procedure at any hospital in Alberta
Sampling Method: Non-Probability Sample
Enrollment: 46000 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevelance of diabetes among surgical population | 11/2019-12/2023
  Determine the incidence of diabetes in the surgical population
HB1AC measuerment in diabetic patients | 11/2019-12/2023
  Determine the incidence of valid HbA1C in diabetic patients presenting for surgery
Long term diabetes control among surgical patients | 11/2019-12/2023
  Determine long-term diabetes control through assessment of HbA1C values in diabetic patients presenting for surgery

SECONDARY OUTCOMES:
In hospital mortality | 11/2019-12/2023
  Determine association between HbA1C and in hospital mortality
Post-operative length of stay | 11/2019-12/2023
  Determine association between HbA1C and post-operative length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The study team still debating sharing the IPD

REFERENCES:
- [Background] Dronge AS, Perkal MF, Kancir S, Concato J, Aslan M, Rosenthal RA. Long-term glycemic control and postoperative infectious complications. Arch Surg. 2006 Apr;141(4):375-80; discussion 380. doi: 10.1001/archsurg.141.4.375. PMID 16618895
- [Background] Jones CE, Graham LA, Morris MS, Richman JS, Hollis RH, Wahl TS, Copeland LA, Burns EA, Itani KMF, Hawn MT. Association Between Preoperative Hemoglobin A1c Levels, Postoperative Hyperglycemia, and Readmissions Following Gastrointestinal Surgery. JAMA Surg. 2017 Nov 1;152(11):1031-1038. doi: 10.1001/jamasurg.2017.2350. PMID 28746706
- [Background] Stryker LS, Abdel MP, Morrey ME, Morrow MM, Kor DJ, Morrey BF. Elevated postoperative blood glucose and preoperative hemoglobin A1C are associated with increased wound complications following total joint arthroplasty. J Bone Joint Surg Am. 2013 May 1;95(9):808-14, S1-2. doi: 10.2106/JBJS.L.00494. PMID 23636187
- [Background] van den Boom W, Schroeder RA, Manning MW, Setji TL, Fiestan GO, Dunson DB. Effect of A1C and Glucose on Postoperative Mortality in Noncardiac and Cardiac Surgeries. Diabetes Care. 2018 Apr;41(4):782-788. doi: 10.2337/dc17-2232. Epub 2018 Feb 13. PMID 29440113

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT06589466/Prot_SAP_000.pdf